CLINICAL TRIAL: NCT04127162
Title: Short-Period Temporal Dispersion Repolarization Markers and In-Hospital Mortality in Decompensated Heart Failure: A Pilot Study
Brief Title: Heart Failure Decompensation And In-Hospital Mortality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Piccirillo, professor, University of Roma La Sapienza
Other Study IDs: CHF_NTproBNP
Record Dates: First submitted 2019-10-13; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Chronic Heart Failure; Decompensated Heart Failure; Morality
Keywords: Temporal Dispersion of Repolarization Phase; proBNP; QTVI; QT; Tpeak-Tend

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- alive
- dead

SUMMARY:
Background and objectives Heart failure is a leading cause of morbidity and mortality worldwide and it is a major cause of emergency department access for cardiovascular disease patients. Aim of this study is to identify the markers, based on short-term temporal repolarization dispersion, capable to individuate decompensated chronic heart failure (CHF) patients at high mortality risk.

Method: We will obtain the following variables from ECG monitor, via mobile phone, during 5-minute recordings in decompensated CHF patients: RR, QT end (QTe), QT peak (QTp) and T peak to T end (Te) and we calculated mean, standard deviation (SD) and normalized index (N).

ELIGIBILITY:
Inclusion Criteria:

* at least one symptom or sign compatible with a decompensation and/or a previous documented history of CHF

Exclusion Criteria:

* pneumonia
* pulmonary embolism

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: decompensated heart failure patients admitted to the emergency department with dyspnea and other clinical signs of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 months
  in-hospital mortality in decompensated heart failure patients

REFERENCES:
- [Derived] Moscucci F, Sciomer S, Maffei S, Meloni A, Lospinuso I, Carnovale M, Corrao A, Di Diego I, Caltabiano C, Mezzadri M, Mattioli AV, Gallina S, Rossi P, Magri D, Piccirillo G. Sex Differences in Repolarization Markers: Telemonitoring for Chronic Heart Failure Patients. J Clin Med. 2023 Jul 16;12(14):4714. doi: 10.3390/jcm12144714. PMID 37510828
- [Derived] Piccirillo G, Moscucci F, Bertani G, Lospinuso I, Sabatino T, Zaccagnini G, Crapanzano D, Diego ID, Corrao A, Rossi P, Magri D. Short-period temporal repolarization dispersion in subjects with atrial fibrillation and decompensated heart failure. Pacing Clin Electrophysiol. 2021 Feb;44(2):327-333. doi: 10.1111/pace.14158. Epub 2021 Jan 12. PMID 33382121
- [Derived] Piccirillo G, Moscucci F, Bertani G, Lospinuso I, Mastropietri F, Fabietti M, Sabatino T, Zaccagnini G, Crapanzano D, Di Diego I, Corrao A, Rossi P, Magri D. Short-Period Temporal Dispersion Repolarization Markers Predict 30-Days Mortality in Decompensated Heart Failure. J Clin Med. 2020 Jun 16;9(6):1879. doi: 10.3390/jcm9061879. PMID 32560151